CLINICAL TRIAL: NCT01219413
Title: The Effect of Aliskiren on Proteinuria in Chronic Nondiabetic Kidney Disease: a Double Blind Cross-over Randomized Controlled Trial
Brief Title: Influence of Aliskiren on Proteinuria
Acronym: ALIPRES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Leszek Tylicki, Prof., Medical University of Gdansk
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ST-4/Aliskiren/01
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Kidney Disease; Proteinuria; Blood Pressure
Keywords: aliskiren; renin inhibitor; proteinuria; chronic kidney diseases; ACE inhibitor
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria | interventions — aliskiren; Perindopril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aliskiren, placebo, perindopril (Experimental)
  Interventions: Drug: Aliskiren, Perindopril
- perindopril, placebo, aliskiren (Experimental)
  Interventions: Drug: Aliskiren, Perindopril

INTERVENTIONS:
Drug: Aliskiren, Perindopril — Rasilez 300 mg Prestarium 10 mg
  Other Names: Rasilez 300 mg; Prestarium 10 mg

SUMMARY:
To evaluate the proteinuria lowering efficacy as well as tolerability and safety of the renin inhibitor aliskiren compared with that of placebo and angiotensin converting enzyme inhibitor perindopril in patients with non-diabetic chronic renal disease.

DETAILED DESCRIPTION:
Proteinuria is a major risk factor for progression to end-stage renal disease in both diabetic and nondiabetic nephropathies. Angiotensin II and aldosterone are the key players in the development of renal failure, either directly by promoting tissue fibrosis or indirectly through their action on glomerular hemodynamic and proteinuria. Therefore, pharmacological inhibition of the renin-angiotensin-aldosterone system (RAAS) may have a beneficial impact on proteinuria and chronic kidney diseases progression. Recently, renin inhibitors, a new class of drugs that selectively inhibits angiotensin II formation at the first step of the RAAS cascade has been introduced to clinical practice. Aliskiren is the first orally bioavailable direct renin inhibitor approved for the treatment of hypertension. Blood pressure (BP)-lowering effect of aliskiren is associated with a decreased generation of angiotensin I, as it blocks its generation from angiotensinogen, by inhibiting the active enzymatic site of renin. The investigators plan this study to evaluate the short-term effects of treatment with aliskiren to those of placebo and ACEI perindopril on proteinuria.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* chronic non-diabetic proteinuric nephropathy
* creatinine clearance above 30 ml/min
* stable proteinuria above 500 mg/ 24 hours
* blood pressure above 125/75 mmHg and below 150/95 mmHg
* no steroids or other immunosuppressive treatment for a minimum of six months before the study

Exclusion Criteria:

* unstable coronary heart disease
* decompensated congestive heart failure in the previous 6 months
* episode of malignant hypertension or stroke in the history
* diabetes
* creatinine clearance below 30 ml/min

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-03; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Investigate the antiproteinuric effect of adding aldosterone antagonist, spironolactone to the combination therapy with angiotensin converting enzyme inhibitor and AT-1 receptor blocker in maximal recommended doses. reduction of proteinuria | march 2014 - april 2014

SECONDARY OUTCOMES:
reduction of blood pressure | march 2013 - april 2014

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Gdansk, Gdansk, Pomeranian Voivodeship, Poland